CLINICAL TRIAL: NCT02660203
Title: Impact of Ipsilateral Decubitus Forced Expiration On Duration of Pleural Drainage After Pulmonary Surgery in Children : Randomized Trial
Brief Title: Impact of Forced Expiration On Pleural Drainage Duration (KPDP)
Acronym: KPDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRIP-14/EC/KPDP; 2015-A01549-40 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-01-05; First posted 2016-01-21 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Malformations; Child
Keywords: chest physiotherapy; post operative period; forced expiration; pleural drainage duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- forced expiration (Experimental): 2 daily sessions of forced expiration on ipsilateral decubitus from day 1 after surgery until chest tube removal
  Interventions: Procedure: Forced expiration
- control (No Intervention): No session of forced expiration

INTERVENTIONS:
Procedure: Forced expiration — Amongst chest physiotherapy technics, forced expiration is one of the passive procedures used in pediatrics.
  The patient is positioned on ipsilateral decubitus and the physiotherapist is behind the patient, placing one hand on the patient abdomen and the other on the patient lateral chest. During expiration, the abdominal hand apply a pressure directed posteriorly and superiorly for the patient. Simultaneously, the thoracic hand apply a pressure posteriorly and inferiorly for the patient. The session's duration is 15 minutes after what the physiotherapist replace the patient in dorsal decubitus.Two sessions a day will be performed
  Arms: forced expiration

SUMMARY:
Following thoracic surgery, pleural effusion in pleural cavity requires post-operative drainage.

Pleural effusion is responsible for pulmonary congestion, atelectasis, hypoventilation, lower efficacy of diaphragmatic curse, lower pulmonary reexpansion and vicious attitude. These complications could be avoided by respiratory physiotherapy.

Forced expiration technic in ipsilateral decubitus is one of these technics but has never been proved better than other technics regarding its efficiency.

The aim of the study is to compare the impact of such a technic on post operative thoracic drainage after pulmonary, pleural or mediastinal pediatric surgery.

DETAILED DESCRIPTION:
Following thoracic surgery, pleural effusion in pleural cavity requires post-operative drainage, most often for few days (2 to 5 days) until fluid quantity is lower than 50 mL / 24h.

Pleural effusion may cause pulmonary congestion, atelectasis, hypoventilation, lower efficacy of diaphragmatic curse, lower pulmonary reexpansion and vicious attitude.

Respiratory physiotherapy in such situations has different aims : pulmonary decongestion and reexpansion, aid for drainage and pleural fluid reduction, avoiding complications and preventing vicious attitudes.

These aims are learned in Physiotherapy formation institutes. The forced expiration technic in ipsilateral decubitus is justified by pleural physiology and is used after pediatric surgery without any scientific evidence regarding his efficacy Using pulmonary physiotherapy after pulmonary, mediastinal or pleural surgery for children is not systematic and depends on prescriber without any professional recommendation.

Actually no scientific evidence regarding technical or postural indicates improvement of effusion drainage.

It seems to be necessary to validate efficiency of such a technic and evaluate its consequences on post-operative pain. Furthermore, this pleural drainage impacts directly the duration of hospitalization and paramedical workload

ELIGIBILITY:
Inclusion Criteria:

* Children 0-4 years
* In front have a mediastinum or lung surgery (lung segmentectomy or lobectomy or non anatomical lung resection) with pleural drainage, regardless of the type drain
* Whose parents or the holder of parental authority have signed a consent
* Whose parents or the holder of parental authority are affiliated to a social security scheme

Exclusion Criteria:

* chest trauma
* Oncology (chest tumors, lung metastases)
* Drained Pleuropneumopathies
* Spine Surgery
* Heart surgery
* Surgery for pectus excavatum
* Route of anterior surgical approach sternotomy chest kind
* Patients intubated and / or ventilated
* Patients with preoperative sepsis

Ages: 1 Day to 48 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
assessment of pleural drainage duration | 3 days
  During the post-operative period until chest tube removal amount of pleural liquid drained is daily assessed.

SECONDARY OUTCOMES:
assessment of total amount of pleural liquid drained | 3 days
  Calculating cumulative volume of liquid provided by the drain (until it reaches 50 cc or less during the last day) during the post-operative period until chest tube removal
Assessment of pain | 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 5, 48
  Pain scale score (EVENDOL 0 to 15)
patient's respiratory parameters | 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48
  level of oxygen dependency (L/min) during the post-operative period until chest tube removal
paramedical workload | 3 days
  Paramedical workload assessed by the time consumption (Hours) due to drainage tube
Oxygen blood saturation | 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48
  Oxygen blood saturation (%) during the post-operative period until chest tube removal

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CHICOISNE, Mrs, Principal Investigator — UH TOURS; Hubert LARDY, MD, Principal Investigator — UH Tours
Locations (10):
- France (10):
  - Uh Angers, Angers
  - UH BREST, Brest
  - Hospices civiles Lyon, Bron
  - UH of PARIS - KREMLIN BICETRE Hospital, Le Kremlin-Bicêtre
  - Uh Limoges, Limoges
  - UH Marseille, Marseille
  - Uh Nantes, Nantes
  - UH of PARIS - NECKER Hospital, Paris
  - UH of PARIS - Robert Debre Hospital, Paris
  - UH Tours, Tours